CLINICAL TRIAL: NCT07059312
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JADE101 Administered Subcutaneously in Healthy Volunteers
Brief Title: A Phase 1 Study of JADE101 in Healthy Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jade Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: JADE101-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: JADE101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JADE101 (Experimental): Subcutaneous (SC) injection of JADE101
  Interventions: Drug: JADE101
- Placebo (Placebo Comparator): Subcutaneous (SC) injection of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JADE101 — JADE101 is supplied as sterile solution to be administered by SC injection.
  Arms: JADE101
Drug: Placebo — Placebo solution to be administered at a matching volume by SC injection.
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of JADE101 compared to placebo in healthy participants.

DETAILED DESCRIPTION:
This is a single center, Phase 1, double-blind, placebo-controlled, randomized, first-in-human (FIH), single ascending dose study evaluating the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of JADE101 in healthy participants. The study will enroll approximately 32 healthy volunteers. JADE101 will be administered by a subcutaneous injection. The results of this study will help inform the dosing and frequency of dosing in future studies of JADE101.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants 18-55 years of age, inclusive
2. A body weight between 50-100 kg and a body mass index (BMI) between 18.0 - 32.0 kg/m2 (all inclusive) at screening
3. Willing and able to comply with the study site stay, scheduled visits, and study procedures
4. Willing and able to comply with using two methods of contraception (one being highly effective) and lifestyle requirements from admission through the end of the study

Exclusion Criteria:

1. Harmful alcohol use
2. Smoking/vaping or heavy tobacco use within 2 years prior to screening
3. Known history of abuse of illicit drugs
4. Nursing, lactating or pregnant, or who have plans to become pregnant during the study
5. Known history of clinically significant disease
6. Known history of immunodeficiency disorder
7. History of clinically significant allergic reactions or hypersensitivity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-08-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Single Ascending Doses of JADE101 in Healthy Participants | Day 1 through 48 weeks
  Incidence of treatment-emergent adverse events

SECONDARY OUTCOMES:
Cmax | Day 1 through 48 weeks
  Maximum observed serum concentration
Tmax | Day 1 through 48 weeks
  Time to reach Cmax
AUClast | Day 1 through 48 weeks
  The area under the concentration-time curve from time zero to the time of the last observed quantifiable (non-zero) concentration
T1/2 | Day 1 through 48 weeks
  Apparent first-order terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, MD, Study Director — Jade Biosciences, Inc.
Locations (1):
- NZCR, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No